CLINICAL TRIAL: NCT05940857
Title: US National OCS Liver Perfusion (OLP) Registry
Acronym: National OLP
Status: Recruiting | Type: Observational
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Other Study IDs: OCS-LIVER-OLP-II
Record Dates: First submitted 2023-06-29; First posted 2023-07-11 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Liver Transplant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- OCS Liver Transplant Recipients: The US National OLP Registry will enroll all liver transplant recipients who are transplanted with an OCS-perfused donor liver in the Registry.
  Interventions: Device: OCS Liver
- Non-OCS Liver Transplant Recipients: Patients transplanted using other preservation modalities for clinical outcomes.

INTERVENTIONS:
Device: OCS Liver — The TransMedics® Organ Care System (OCS) Liver is an FDA approved portable extracorporeal liver perfusion and monitoring system.
  Groups: OCS Liver Transplant Recipients

SUMMARY:
This Registry is a sponsor-initiated, multi-center, observational, post-approval registry with an independent academic oversight.

TransMedics has contracted with United Network for Organ Sharing (UNOS) the Federal manager of the U.S. national transplant outcomes registry to obtain data that is routinely collected by the Organ Procurement and Transplantation Network (OPTN) on all transplanted organs in the U.S. for both the OCS liver transplanted patients as well as patients transplanted using other preservation modalities. Additional data will be collected by participating centers using OCS Liver perfusion.

ELIGIBILITY:
All liver transplant recipients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All liver transplant recipients who are transplanted with an OCS-perfused donor liver will be enrolled in the Registry. Patients' clinical outcomes will be followed until the later of 5 years post-transplant, loss to follow-up or death.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2021-10-14 (Actual); Primary Completion 2031-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Survival | 5 years post-transplant
  Recipients' patient and graft survival rates will be the primary clinical outcomes measures for all OCS Liver transplanted recipients compared to recipients receiving liver transplants using non-OCS preservation methods (cold static storage or other perfusion devices or a combination of both). This data will be obtained directly from UNOS/OPTN database.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elbetanony, MD, Study Director — TransMedics
Locations (22):
- United States (22):
  - University of Alabama, Birmingham, Alabama
  - Mayo Clinic Hospital Arizona, Phoenix, Arizona
  - University of California San Diego, La Jolla, California
  - University of California San Francisco, San Francisco, California
  - Mayo Clinic Hospital Florida, Jacksonville, Florida
  - Emory University Hospital, Atlanta, Georgia
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic Hospital Minnesota, Rochester, Minnesota
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - NY Presbyterian Hospital/Columbia Univ. Medical Center, New York, New York
  - Carolinas Medical Center/Atrium Health, Charlotte, North Carolina
  - Duke Medical Center, Durham, North Carolina
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Houston Methodist, Houston, Texas
  - University Hospital, University of Texas Health Science Center, San Antonio, Texas
  - University of Utah Medical Center, Salt Lake City, Utah